CLINICAL TRIAL: NCT04241874
Title: Effects of Positive End-expiratory Pressure With and Without Inspiratory Synchronization During Moderate to Severe ARDS
Brief Title: PEEP and Spontaneous Breathing During ARDS
Acronym: EARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EARDS
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low PEEP and full inspiratory synchronization (Experimental): PEEP = 5 cmH2O + clinically selected pressure support (PSVclin)
  Interventions: Other: Mechanical Ventilation
- High PEEP and full inspiratory synchronization (Experimental): PEEP = 15 cmH2O + clinically selected pressure support (PSVclin)
  Interventions: Other: Mechanical Ventilation
- Low PEEP and inspiratory desynchronization (Experimental): PEEP = 5 cmH2O + bilevel positive airway pressure (Respiratory rate 15 breaths/minute, inspiratory time=1 sec, Inspiratory pressure=PSVclin+PEEP, PS=0 cmH2O)
  Interventions: Other: Mechanical Ventilation
- High PEEP and inspiratory desynchronization (Experimental): PEEP = 15 cmH2O + bilevel positive airway pressure (Respiratory rate 15 breaths/minute, inspiratory time=1 sec, Inspiratory pressure=PSVclin+PEEP, PS=0 cmH2O)
  Interventions: Other: Mechanical Ventilation

INTERVENTIONS:
Other: Mechanical Ventilation — Respiratory support through mechanical ventilator

SUMMARY:
Prospective, physiological study to systematically assess the effects of high positive end-expiratory pressure (PEEP) with and without inspiratory synchronization in patients with moderate to severe acute respiratory distress syndrome (ARDS) exhibiting intense inspiratory effort while on assisted ventilation.

DETAILED DESCRIPTION:
This prospective, physiological, randomized, cross-over study will be conducted in the 20-bed general ICU of the Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy. Patients with ARDS will be screened for eligibility. ARDS will be defined according to the Berlin Definition.

Intubated patients fulfilling ARDS criteria, undergoing assisted ventilation as per clinical decision and exhibiting intense inspiratory effort (occlusion pressure equal or greater than 13 cmH2O) will be enrolled.

Patients will be placed in a 30°-45° head up position during all study phases. According to our institution protocol, pressure support setting will be selected by the attending physician to target a predefined tidal volume range of 6-8 mL/kg of predicted body weight (PBW) (female PBW [kg] = 45.5 + 0.91 [cm of height - 152.4]; male PBW [kg] = 50 + 0.91 [cm of height - 152.4]).The lowest pressure support level allowed will be 7 cmH2O, even if Vt <8 ml/Kg PBW is not achieved.

In each patient, four different ventilator settings will be applied in a random order. Each step will last 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* (a) ARDS according to the Berlin definition (ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) ≤ 300 mmHg);
* (b) assisted ventilation, as prescribed by the attending physician
* (c) intense inspiratory effort, defined as a negative deflection in the airway pressure equal or greater than 13 cmH2O in the first breath recorded during an end-expiratory occlusion

Exclusion Criteria:

Pregnancy, clinically documented barotrauma, contraindication to electrical impedance tomography (EIT) use (e.g., presence of pacemaker or automatic implantable cardioverter defibrillator), impossibility to place the EIT belt in the right position (e.g., presence of surgical wounds dressing), and any contraindication to the insertion of a nasogastric tube (eg, recent upper-gastrointestinal surgery, esophageal varices), chest tubes with active air leaks, fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Inspiratory effort | 45 minutes
  The negative deflection in esophageal pressure during inspiration

SECONDARY OUTCOMES:
Oxygenation | 45 minutes
  Ratio of PaO2 to FiO2
Respiratory mechanics | 45 minutes
  Respiratory mechanics assessed by end-inspiratory occlusion
Lung mechanics | 45 minutes
  Respiratory mechanics assessed by esophageal pressure monitoring during an end-inspiratory occlusion
Work of breathing | 45 minutes
  Esopghageal pressure pressure-time product per minute
Respiratory rate | 45 minutes
  Respiratory rate per minute
Regional Tidal volume distribution | 45 minutes
  Distribution of tidal volume in the different lung zones, assessed by electrical impedance tomography
Alveolar recruitment | 45 minutes
  Change in end-expiratory lung impedance, assessed by electrical impedance tomography
Pendelluft | 45 minutes
  Occurrence of intra-tidal shift of gas within different lung regions at beginning of inspiration
Carbon dioxide | 45 minutes
  Blood carbon dioxide, as assessed by arterial blood gas analysis
Tidal volume | 45 minutes
  Average Tidal volume received by the patient
Dynamic transpulmonary driving pressure | 45 minutes
  The average positive swing in transpulmonary driving pressure during tidal breathing

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Bello, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS; Massimo Antonelli, MD, Study Director — Fondazione Policlinico A. Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be made available upon a reasonable request

REFERENCES:
- [Derived] Bello G, Giammatteo V, Bisanti A, Delle Cese L, Rosa T, Menga LS, Montini L, Michi T, Spinazzola G, De Pascale G, Pennisi MA, Ribeiro De Santis Santiago R, Berra L, Antonelli M, Grieco DL. High vs Low PEEP in Patients With ARDS Exhibiting Intense Inspiratory Effort During Assisted Ventilation: A Randomized Crossover Trial. Chest. 2024 Jun;165(6):1392-1405. doi: 10.1016/j.chest.2024.01.040. Epub 2024 Jan 29. PMID 38295949